CLINICAL TRIAL: NCT03886584
Title: Source Monitoring Déficit in Neuropsychiatric Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A00584-51
Record Dates: First submitted 2019-03-11; First posted 2019-03-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Psychiatric Disorder
Keywords: Bipolar Disorder; Source-monitoring
MeSH Terms: conditions — Mental Disorders; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: 2 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with with neuropsychiatric conditions (Experimental): In this arm, five groups :
  * Patients with DFT, diagnosed according Racovsky criteria
  * Patients with Lewi Body dementia, diagnosed according McKeith criteria
  * Patients with pre-demential Alzheimer, diagnosed according Dubois criteria
  * Patients with Alzheimer, diagnosed according MMSE
  * Patients with bipolar disorder, diagnosed according DSM 5
  Interventions: Other: Monitoring source test
- Healthy subjects (Active Comparator): Healthy controls appaired in age, sex and educational level
  Interventions: Other: Monitoring source test

INTERVENTIONS:
Other: Monitoring source test — Internal- and external-monitoring correct responses and inversions

SUMMARY:
the investigators will measure source-monitoring ability in patients with several neuropsychiatric condition and in healthy controls appaired in age, sex and educational level. Source-monitoring will be measured thanks to internal- and reality-monitoring informatic tasks.The investigators hypothesized patients with fronto-temporal abnormalities would show more marked deficits than patients with only frontal abnormalities.

DETAILED DESCRIPTION:
Source-monitoring abilities will be measured thanks to reality-monitoring testing (i.e. the ability to distinguish internal-generated events from external ones) and internal-monitoring testing (i.e. the ability to distinguish an imagined source from a performed one). A source-monitoring deficit have been demonstrated in patients with psychiatric conditions such as schizophrenia and seems linked to frontotemporal abnormalities (frontotemporal dysconnectivity and temporal hypoactivity). With a total of 150 patients, the investigators will include 30 patients per group: patients with pre-dementia stage Alzheimer, Alzheimer, Fronto-Temporal dementia, Lewy Body dementia or Parkinson and Bipolar Disorder, with the hypothesis that Bipolar Disorder patients will present less marked deficit. The investigators will recruit 150 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who gave their free and informed consent;
* Men and women;
* Aged 18 to 80;
* Having normal or corrected vision;
* Mastering the French language (read and spoken);
* All subjects will not have a working memory deficit preventing the test from being passed (MMSE short version):AM patients should have a score of <MMSE <26; Patients with pre-dementia AD will be diagnosed according to Dubois criteria (Dubois et al., 2016); patients with early FTD will be diagnosed according to Rascovsky's criteria (Rascovsky et al., 2011); Patients with DCL will be diagnosed according to McKeith's criteria (McKeith et al., 2005), TBP patients will be diagnosed using DSM 5 criteria (Arlington VA, 2013).

Exclusion Criteria:

* Inadmissibility of the consent or refusal of the subject.
* Patients under guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
measure source memory performance | one year
  in patients with neuropsychiatric disorders with or without temporal involvement (pre-dementia Alzheimer's disease, Alzheimer's disease - AD, fronto-temporal dementia - DFT, Lewy body dementia - DCL and bipolar disorder - TBP) and healthy volunteers matched in age, gender, and level of education.

SECONDARY OUTCOMES:
measure the recognition of distractors | one year
  words not presented during the source monitoring test phase but presented during the recall phase. This measure will allow us to avoid that a disturbance invading the working memory or attentional capacities does not compromise the good realization of the task.

CONTACTS AND LOCATIONS:
Overall Officials: JEROME BRUNELIN, PHD, Principal Investigator — Centre Hospitalier Le Vinatier - CRNL - INSERM
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No